CLINICAL TRIAL: NCT02189993
Title: Limited Long Term Survival in Patients After In-hospital Intestinal Failure Requiring Total Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Leendert Oterdoom, Dr., Amsterdam UMC, location VUmc
Other Study IDs: TPN-01
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Nutrition Disorders
Keywords: Mortality; Long term follow-up; Parenteral Nutrition, Total
MeSH Terms: conditions — Nutrition Disorders; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Parenteral Nutrition Use: The cohort investigated consisted of patients with intestinal failure requiring total parenteral nutrition use.

SUMMARY:
The purpose of this study is to determine what the long term survival is after in hospital use of total parenteral nutrition due to intestinal failure.

Earlier studies only followed patients for a maximum of 6 months or included only very specific patients. We were interested in all patients in our hospital and followed them for up to 2 years.

DETAILED DESCRIPTION:
Extensive description is not desired

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients on TPN

Exclusion Criteria:

* patients from the Pediatric and Haematological Departments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring total parenteral nutrition during in hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Up to 1427 days

CONTACTS AND LOCATIONS:
Overall Officials: Leendert Oterdoom, MD PhD, Principal Investigator — VUMC
Locations (1):
- Department of Gastroenterology and Hepatology, Small Bowel Unit, VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Oterdoom LH, Ten Dam SM, de Groot SD, Arjaans W, van Bodegraven AA. Limited long-term survival after in-hospital intestinal failure requiring total parenteral nutrition. Am J Clin Nutr. 2014 Oct;100(4):1102-7. doi: 10.3945/ajcn.114.087015. Epub 2014 Aug 13. PMID 25240075